CLINICAL TRIAL: NCT02263716
Title: Actigraphy to MEasuRe Intensive Care Unit Activity (AMERICA)
Brief Title: Actigraphy to MEasuRe Intensive Care Unit Activity
Acronym: AMERICA
Status: Completed | Type: Observational
Sponsor: Vanderbilt University (Other)
Responsible Party: Principal Investigator, Nathan Brummel, Instructor in Medicine, Vanderbilt University
Organization: Vanderbilt University Medical Center (Other)
Other Study IDs: 141504
Record Dates: First submitted 2014-10-02; First posted 2014-10-13 (Estimated); Last update posted 2017-01-06 (Estimated); Status verified 2017-01

CONDITIONS: Disability; Physical Activity; Aging; Critical Illness
Keywords: Physical Activity; Intensive Care; Activities of Daily Living; Delirium; Sepsis; Mechanical Ventilation; Critical Care; Critical Illness; Aging; Accelerometery
MeSH Terms: conditions — Motor Activity; Critical Illness; Delirium; Sepsis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Accelerometer: Utilize accelerometers to measure activity in a diverse population of patients with medical or surgical critical illness.

SUMMARY:
This study is to determine whether accelerometry can be used to measure physical activity occurring during routine clinical care in a diverse population of patients with medical or surgical critical illness.

DETAILED DESCRIPTION:
Patients that meet inclusion criteria will have a wristwatch size, lightweight ActiGraph GT3X+ placed at each of three body sites, the dominant-side wrist, right hip and dominant-side ankle to objectively measure physical activity. Patients will wear the ActiGraph devices during two 30-minute periods of direct observation. To compare activity counts measured by the ActiGraph devices with directly observed purposeful physical activity, we will record the time and type of physical activity performed by patients such as sitting at the edge of the bed, sitting in a bedside chair, transferring to a chair, standing and ambulating. The data acquired from this observational (AMERCIA) study will seek to establish the feasibility of using accelerometers to measure activity in a diverse population of patients with medical or surgical critical illness.

ELIGIBILITY:
Inclusion Criteria:

Patients will be included if they are:

1. adult patients,
2. admitted to the medical or surgical ICU,
3. receiving or have received invasive or non-invasive mechanical ventilation for respiratory failure or vasopressors for shock (i.e., cardiogenic, hemorrhagic, septic or undifferentiated shock) within the last 48 hours, and
4. who are receiving routine physical and occupational therapy.

Exclusion Criteria:

Patients will be excluded if they meet any of the following criteria:

1. Those who have severe physical disability that prevented independent living prior to their illness,
2. Those unable to speak and communicate in English,
3. Expected death within 24 hours of enrollment or lack of commitment to aggressive treatment by the family or medical team (i.e., likely to withdraw life support measures within 24 hours of screening),
4. Inability to obtain informed consent from authorized surrogate;

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: A diverse population of adult patients with medical or surgical critical illness in the ICU.
Sampling Method: Non-Probability Sample
Enrollment: 25 (Actual)
Dates: Start 2015-07; Primary Completion 2016-01 (Actual); Study Completion 2016-02 (Actual)

PRIMARY OUTCOMES:
Feasibility of accelerometers to measure physical activity in patients with a critical illness. | 1 Day
  To determine the validity of activity counts from each of the three accelerometry sites (wrist, hip and ankle) with direct observation acting as the reference.

SECONDARY OUTCOMES:
Tolerability of accelerometry devices. | 1 Day
  We will assess tolerability of the ActiGraph devices through the assessment of the number of total hours devices are worn (out of 120 hours of possible measurement time). We will record the time of device removal and replacement as well as reasons for device removal. Patients will be routinely evaluated for device-related discomfort and devices will be repositioned or removed accordingly. Finally, at the conclusion of the study period, patients will be surveyed regarding the tolerability of the devices.

CONTACTS AND LOCATIONS:
Overall Officials: Nathan E. Brummel, MD, Principal Investigator — Vanderbilt University Medical Center
Locations (1):
- Vanderbilt University Medical Center, Nashville, Tennessee, United States